CLINICAL TRIAL: NCT00017732
Title: Carrier Frequency and Incidence of Smith-Lemli-Opitz Syndrome in African Americans
Brief Title: Estimation of the Carrier Frequency and Incidence of Smith-Lemli-Opitz Syndrome in African Americans
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010191; 01-CH-0191
Record Dates: First submitted 2001-06-08; First posted 2001-06-11 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-03

CONDITIONS: Smith-Lemli-Opitz Syndrome
Keywords: Malformations; Ethnicity; Mutations; Cholesterol; Metabolism; Smith-Lemli-Opitz Syndrome; SLOS; Cholesterol Metabolism
MeSH Terms: conditions — Smith-Lemli-Opitz Syndrome

SUMMARY:
RSH/Smith-Lemli-Opitz syndrome (SLOS) is one that causes mental retardation. It is common in the Caucasian population but rare in African American and African black populations. It has been shown that SLOS is caused by a specific defect in DHCR7, an enzyme used in cholesterol metabolism. Studies have already been done to determine the frequency of the SLOS-causing mutations in various geographic Caucasian populations. This study will investigate the frequency of the DHCR7 mutations in the African American population. If the frequency observed suggests that SLOS cases are not being identified in this ethnic group, the study will provide the rationale for future studies to identify these patients.

The sample size will be 1,600. The study population will consist of archived biological specimens in the form of newborn screening blood spots from two newborn screening centers, one in Maryland and one in Pennsylvania. Subjects will be of African American ethnicity, including blacks of African, Caribbean, and Central American descent.

Genomic DNA will be extracted from blood spots and screened for the six common SLOS mutations. If SLOS syndrome is found, followup will be attempted for the Maryland samples (the Pennsylvania samples will be totally anonymous).

DETAILED DESCRIPTION:
RSH/Smith-Lemli-Opitz syndrome (SLOS) is a multiple congenital anomaly/mental retardation syndrome caused by inborn error of cholesterol metabolism (Tint et al. 1994; Opitz 1999; Kelley 2000). Recent studies have shown SLOS to be one of the most common inherited metabolic defects in the Caucasian population. SLOS is believed to be rare in people of Chinese, Japanese, Indian, and Korean origin as well as in the African American and African Black population (Tsukahara et al. 1998; Yu et al 2000a; Witsch-Baumgartner et al. 2000; Witsch-Baumgartner et al. 2001, Battaile et al. 2001). The frequency spectra of DHCR7 mutations have been established for American Caucasians (Yu et al. 2000b, Battaile et al. 2001), mixed American Caucasian collection of patients (Witsch-Baumgartner et al 2000), for European ethnic groups from Poland, German/Austria, Great Britain (Witsch-Baumgartner et al. 2001) and from Italy (De Brasi et al. 1999). In these Caucasian populations, the most common mutations (IVS8-1G>C, W151X, V326L, R352W, R404C and T93M) account for 60% of SLOS mutant alleles. These suggest that frequent SLOS-causing mutations have different geographic origins and histories. This project will investigate the frequency gradient of DHCR7 mutations in the African American population.

ELIGIBILITY:
INCLUSION CRITERIA:

These will be newborn screening blood spots from African American babies. Samples from Blacks of African, Caribbean and Central American descent will be included. The classification of the infants will be based on the maternal identification as Black or African American by blood spot submission card.

EXCLUSION CRITERIA:

Newborn screening blood spots from non-African American or non-Black babies.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000
Dates: Start 2001-06; Study Completion 2003-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Child Health and Human Development (NICHD), Bethesda, Maryland, United States

REFERENCES:
- [Background] Bzduch V, Behulova D, Skodova J. Incidence of Smith-Lemli-Opitz syndrome in Slovakia. Am J Med Genet. 2000 Jan 31;90(3):260. doi: 10.1002/(sici)1096-8628(20000131)90:33.3.co;2-i. No abstract available. PMID 10678669
- [Background] Battaile KP, Battaile BC, Merkens LS, Maslen CL, Steiner RD. Carrier frequency of the common mutation IVS8-1G>C in DHCR7 and estimate of the expected incidence of Smith-Lemli-Opitz syndrome. Mol Genet Metab. 2001 Jan;72(1):67-71. doi: 10.1006/mgme.2000.3103. PMID 11161831
- [Background] Angle B, Tint GS, Yacoub OA, Clark AL. Atypical case of Smith-Lemli-Opitz syndrome: implications for diagnosis. Am J Med Genet. 1998 Dec 4;80(4):322-6. PMID 9856557